CLINICAL TRIAL: NCT06644495
Title: Post-Market Surveillance Study of ALK-Positive Advanced NSCLC Participants Treated With Iruplinalkib
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRU-PMS-001
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the safety and efficacy of participants diagnosed with anaplastic lymphoma kinase (ALK)-positive advanced non-small cell lung cancer (NSCLC) who are being treated with Iruplinalkib or planned to receive Iruplinalkib treatment in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed patients with locally-advanced or metastatic ALK-positive non-small cell lung cancer.
* Currently receiving, or planned to receive treatment with Iruplinalkib.
* Subjects had imaging reports of chest and abdominal enhanced CT and brain MRI within 42 days prior to the first dose of Iruplinalkib as 1L treatment for locally-advanced or metastatic ALK-positive non-small cell lung cancer.
* Subjects had routine and biochemical reports within 30 days prior to the first dose of Iruplinalkib as 1L treatment for locally-advanced or metastatic ALK-positive non-small cell lung cancer.

Exclusion Criteria:

* Patients who had previously been treated with ALK-TKI, but who had previously only been treated with ALK-TKI as neoadjuvant and/or adjunctive treatment could be enrolled.
* Mental disorder or inability to cooperate with examination or follow-up.
* Women known to be pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALK-positive advanced non-small cell lung cancer patients who are being treated with Iruplinalkib or planned to receive Iruplinalkib.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse drug reactions in the overall population | At enrollment and every 3 months thereafter (up to 3 years)

SECONDARY OUTCOMES:
The incidence of greater than or equal to grade 3 AEs, SAEs, AEs resulting in dose reduction/interruption/discontinuation, AESIs, and AEs resulting in death in the overall population | At enrollment and every 3 months thereafter (up to 3 years)
Real-world progression-free survival (rwPFS) for 1L treatment with Iruplinalkib | From the first administration of Iruplinalkib to the date of first documentation of disease progression, or death due to any cause, whichever occurs first (up to 3 years).
Time to treatment failure (TTF) for 1L treatment with Iruplinalkib | From the first administration of Iruplinalkib to the date of first documentation of discontinuation of Iruplinalkib due to any cause (up to 3 years).
Event to first follow-up treatment or death (TFST) for 1L treatment with Iruplinalkib | From the first administration of Iruplinalkib to the date of first documentation of initiation of next line of treatment, or death due to any cause, whichever occurs first (up to 3 years).